CLINICAL TRIAL: NCT05686330
Title: Enhanced Detection and Quickened Diagnosis of Atrial Fibrillation Using the Apple Watch: A Randomised Controlled Trial (EQUAL Study)
Brief Title: Detection and Quantification of Atrial Fibrillation in High-risk Patients Using a Smartwatch Wearable (Apple Watch)
Acronym: EQUAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amsterdam University Medical Centers (UMC), Location Academic Medical Center (AMC) (Other)
Responsible Party: Principal Investigator, Prof. Dr. Arthur A. M. Wilde, Prof. Dr., Amsterdam University Medical Centers (UMC), Location Academic Medical Center (AMC)
Organization: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021_209
Record Dates: First submitted 2022-12-16; First posted 2023-01-17 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation; Cardiac arrhythmia; Smartwatch; Wearable technology; Digital health; Photoplethysmography; Electrocardiography; Remote monitoring; Screening; Randomized controlled trial; Outpatient care; Telemedicine
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Interventional group (Apple watch) (Experimental): These participants will wear a smartwatch (Apple Watch) for 6 months during 12 hours a day. The smartwatch will alarm the participant if an irregular heart rhythm is detected. When a participant experiences any symptoms or receives an irregular heartbeat notification, they can record an ECG with the smartwatch. The ECG will automatically be sent to the Telecure team for evaluation.
  Interventions: Device: Apple Watch
- Control group (No Intervention): Patients in the control group received standard care, which could include conventional rhythm monitoring methods such as Holter monitoring, in-hospital telemetry, or the use of handheld mobile ECG devices, at the discretion of the treating cardiologist. At the end of the study period the investigator will either call the participant to check for these outcome measures.

INTERVENTIONS:
Device: Apple Watch — Smartwatch for detecting atrial fibrillation using photoplethysmography (PPG)
  Other Names: Smartwatch
  Arms: Interventional group (Apple watch)

SUMMARY:
This is a randomized controlled trial evaluating atrial fibrillation (AF) detection through smartwatch-based screening in high-risk patients using an Apple Watch with integrated PPG and ECG functions.

DETAILED DESCRIPTION:
This is a multicenter randomized controlled trial evaluating whether six months of heart rate and rhythm monitoring with a smartwatch (Apple Watch Series 5 or 8) equipped with photoplethysmography (PPG) and ECG functions increases atrial fibrillation (AF) detection in high-risk cardiac patients (age ≥65, CHA₂DS₂-VASc ≥2 for men, ≥3 for women) without previously known AF.

Patients are randomized to either smartwatch-based monitoring or standard care. Participants in the intervention group receive an Apple Watch paired with a smartphone app and are instructed to wear the device for at least 12 hours per day. Continuous rhythm monitoring is performed using PPG, with ECGs recorded upon symptom onset or irregular rhythm detection. ECG data are transmitted via the app to a secure platform and reviewed within 24 hours by an independent eHealth team supervised by a cardiologist. Patients and their treating physicians are notified upon new AF diagnoses.

To evaluate the primary endpoint, a total of 218 patients per arm were required according to the sample size calculation.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65 years
* Chadsvasc score ≥2 for men and ≥ for women at the time of eligibility screening
* Written informed consent as documented by signature from the participant
* Possession of iPhone (6S or later)

Exclusion Criteria:

* Diagnosis of atrial fibrillation or atrial flutter
* Currently on anticoagulation therapy
* Cardiac implanted electronic device (pacemaker, ICD)
* Smartwatch cannot be worn due to comprehensible reasons (allergic reactions, wounds, amputations, other)
* Significant mental or cognitive impairment

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 436 (Actual)
Dates: Start 2022-11-16 (Actual); Primary Completion 2025-07-17 (Actual); Study Completion 2025-07-17 (Actual)

PRIMARY OUTCOMES:
The incidence of atrial fibrillation | 6 months
  Detected with an Apple watch or with any other device such as a holter or on an ECG or telemetry

SECONDARY OUTCOMES:
The time until atrial fibrillation is first detected (days) | 6 months
  The number of days between the date of inclusion and the date AF is detected
The number of patients for whom medication for AF is initiated at the end of the study (anticoagulation and antiarrhythmic drugs) | 6 months
The number of patients that undergo major cardiovascular events during the study period | 6 months
Number of emergency department visits | 6 months
  Emergency department visits that take place during the study period, for any reason
The number of new arrhythmia diagnoses other than AF in each study arm | 6 months
  Detected by either the Apple watch, telemetry, holter or other devices used to detect arrhythmias

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - Cardiology Center of the Netherlands, Amsterdam, North Holland
  - Spaarne Gasthuis, Haarlem, North Holland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] van Steijn NJ, Blommestijn IS, Blok S, Pepplinkhuizen S, Somsen GA, Knops RE, Breukel L, Tijssen JGP, Tulevski II, Croon PM, Winter MM. Enhanced Detection and Prompt Diagnosis of Atrial Fibrillation Using Apple Watch: A Randomized Controlled Trial. J Am Coll Cardiol. 2026 Jan 22:S0735-1097(25)10337-9. doi: 10.1016/j.jacc.2025.11.032. Online ahead of print. PMID 41569211